CLINICAL TRIAL: NCT00003462
Title: Phase I Study of Intrathecal Spartaject-Busulfan in Patients With Neoplastic Meningitis
Brief Title: Intrathecal Busulfan in Treating Patients With Recurrent, Refractory, or Metastatic Leptomeningeal Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0672; DUMC-0672-03-3R5; DUMC-000672-02-3R4; DUMC-000672-00-3R2; DUMC-000672-01-3R3; DUMC-0631-99-4RI; DUMC-625-98-4; DUMC-98045; DUMC-FDR001519; NCI-G98-1463; CDR0000066494 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: leptomeningeal metastases
MeSH Terms: conditions — Central Nervous System Neoplasms; Meningeal Carcinomatosis | interventions — Busulfan

INTERVENTIONS:
Drug: busulfan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving drugs into the thin space between the lining of the spinal cord and brain may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of intrathecal busulfan in treating patients with recurrent, refractory, or metastatic leptomeningeal tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of intrathecal busulfan by a limited escalation dosage schedule in patients with recurrent or refractory leptomeningeal tumors.
* Determine the cerebrospinal fluid and serum pharmacokinetics of busulfan administered via intralumbar or intraventricular routes in these patients.

OUTLINE: This is dose-escalation study.

Patients receive intrathecal busulfan via intralumbar or intraventricular routes twice a week for 2 weeks (4 treatments). Any patient with objective or significant clinical response may continue treatment by receiving the same dose once a week for 2 consecutive weeks, once a week every other week for 3 weeks (2 treatments), and then once a month thereafter until disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of intrathecal busulfan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 12 weeks for 1 year or until disease progression.

PROJECTED ACCRUAL: A total of 5-20 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed neoplasm that is metastatic in the cerebrospinal fluid or leptomeningeal/subarachnoid space

  * Cytologic diagnosis of malignancy in the cerebrospinal fluid or neuroimaging evidence of leptomeningeal tumor by MRI
* Must have a recurrent or refractory leptomeningeal tumor

  * Leptomeningeal tumors of leukemia, lymphoma, and all germ cell tumors must have also failed initial treatment or be recurrent
* No evidence of obstructive hydrocephalus or complete block of the spinal cerebrospinal fluid pathways on prestudy technetium Tc 99m albumin or indium In 111 DTPA flow study

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 8 weeks

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 2.5 mg/dL
* SGOT or SGPT less than 1.5 times normal

Renal:

* BUN less than 30 mg/dL
* Creatinine less than 1.5 mg/dL
* Calcium within normal limits

Neurological:

* Neurological examination stable
* No rapidly progressing or deteriorating neurological deficits

Other:

* No active infectious process
* Magnesium, phosphorus, potassium, chloride, and bicarbonate normal
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy

Chemotherapy:

* At least 6 weeks since prior nitrosoureas or mitomycin
* At least 4 weeks since any other prior chemotherapy
* At least 3 weeks since prior intrathecal chemotherapy
* No other concurrent intrathecal chemotherapy

Endocrine therapy:

* For patients on corticosteroids:

  * Must be on a stable dose of corticosteroids for at least 1 week

Radiotherapy:

* At least 3 weeks since prior radiotherapy to the CNS
* At least 4 weeks since any other prior radiotherapy
* No concurrent radiotherapy to the CNS

Surgery:

* At least 3 weeks since prior surgery

Other:

* No concurrent medication that may interfere with study results (e.g., immunosuppressive agents other than corticosteroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1998-04; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States